CLINICAL TRIAL: NCT00822731
Title: Development of a Predictive Model for Treatment Outcome and Treatment-related Morbidity in a Prospective Cohort Study of Patients With Lymphoma
Brief Title: Samsung Medical Center-Lymphoma Cohort Study
Acronym: SMC-LCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kim, Seok Jin, Associate Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2008-08-068
Record Dates: First submitted 2008-12-30; First posted 2009-01-14 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: Lymphoma; prognosis; morbidity
MeSH Terms: conditions — Lymphoma | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lymphoma (Experimental): patients diagnosed as lymphoma
  Interventions: Drug: Chemotherapy with or without radiotherapy

INTERVENTIONS:
Drug: Chemotherapy with or without radiotherapy — Treatment regimen will be determined by the sub-type of lymphoma
  Other Names: Chemotherapy:CHOP, RCHOP, (R)HyperCVAD

SUMMARY:
The purpose of this study is to establish a model which can predict the treatment outcome and the risk of treatment-related morbidity in patients with lymphoma.

DETAILED DESCRIPTION:
Although the cure rate of lymphoma has been increased due to the development of newer effective drugs, a substantial portion of patients is still suffered from relapse. Furthermore, the treatment-related morbidity is another factor which can make the treatment outcome worse in patients with lymphoma, especially elderly patients. Thus, this study is going to assess following factors which amy probably affect the treatment outcome and the risk of treatment-related morbidity.

1. Biologic factors associated with the aggressiveness of lymphoma

   * molecular markers in serum, cytogenetic markers
2. Factors associated with the risk of treatment-related morbidity

   * comorbidity, nutrition status, performance status, quality of life at diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as lymphoma
* Over 15 years old
* Patients who agreed the enrollment of study
* Informed consent for sampling

Exclusion Criteria:

* Patients who do not want to join the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 953 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 5 years

SECONDARY OUTCOMES:
Treatment response | after completion of primary therapy
Rate of occurrence of toxicity | 2 years from the start of the 1st therapy
Treatment-related morbidity | within 60 days from the previous therapy

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho I, Lee H, Yoon SE, Ryu KJ, Ko YH, Kim WS, Kim SJ. Serum levels of soluble programmed death-ligand 1 (sPD-L1) in patients with primary central nervous system diffuse large B-cell lymphoma. BMC Cancer. 2020 Feb 13;20(1):120. doi: 10.1186/s12885-020-6612-2. PMID 32054467
- [Derived] Kim SJ, Hong M, Do IG, Lee SH, Ryu KJ, Yoo HY, Hong JY, Ko YH, Kim WS. Serum survivin and vascular endothelial growth factor in extranodal NK/T-cell lymphoma, nasal type: implications for a potential new prognostic indicator. Haematologica. 2015 Mar;100(3):e106-9. doi: 10.3324/haematol.2014.116087. Epub 2014 Dec 5. No abstract available. PMID 25480498
- [Derived] Hong JY, Yoon DH, Suh C, Huh J, Do IG, Sohn I, Jo J, Jung SH, Hong ME, Yoon H, Ko YH, Kim SJ, Kim WS. EBV-positive diffuse large B-cell lymphoma in young adults: is this a distinct disease entity? Ann Oncol. 2015 Mar;26(3):548-55. doi: 10.1093/annonc/mdu556. Epub 2014 Dec 4. PMID 25475080
- [Derived] Jung HA, Park S, Cho JH, Kim S, Ko YH, Kim SJ, Kim WS. Prognostic relevance of pretreatment quality of life in diffuse large B-cell lymphoma patients treated with rituximab-CHOP: results from a prospective cohort study. Ann Hematol. 2012 Nov;91(11):1747-56. doi: 10.1007/s00277-012-1516-0. Epub 2012 Jun 28. PMID 22739576